CLINICAL TRIAL: NCT01742130
Title: Early Hydration in Acute Myocardial Infarction: Sodium Bicarbonate Versus Saline for the Prevention on Contrast-induced Acute Kidney Injury
Brief Title: Early Hydration in Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, Medical Doctor, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prato0705
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Contrast Induced Acute Kidney Injury
Keywords: Contrast-induced nephropathy; Contrast media; Angiography; Coronary percutaneous intervention
MeSH Terms: interventions — Glucose; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate (Experimental): Sodium Bicarbonate (154 mEq/L in dextrose and H2O) 3 mL/kg for 1 hour before contrast medium, followed by an infusion of 1 mL/kg/h for 12 hours after the procedure
  Interventions: Drug: sodium bicarbonate solution
- Saline (Active Comparator): Sodium Saline 3 mL/kg for 1 hour before contrast medium, followed by an infusion of 1 mL/kg/h for 12 hours after the procedure
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: sodium bicarbonate solution
  Other Names: 154 mEq/L in dextrose and H2O
  Arms: Sodium bicarbonate
Drug: Isotonic saline
  Other Names: 0.9% sodium chloride
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether hydration with sodium bicarbonate is more effective than hydration with sodium chloride to prevent contrast nephropathy in patients undergoing primary coronary intervention for acute ST elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with AMI candidates for primary PCI presenting within 12 h of symptom onset with ST-segment elevation of more 1 mm in at least two contiguous leads of electrocardiogram.

Exclusion Criteria:

* contrast medium administration within the 10 days
* end-stage renal failure requiring dialysis
* refusal to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast-induced acute kidney injury | 2 days
  contrast-induced acute kidney injury is defined as an increase in serum creatinine >= 0.3 mg/dL over the baseline value within 2 days after the administration of the contrast medium

SECONDARY OUTCOMES:
adverse clinical events | 1 month
  adverse clinical events within 1 month including in-hospital death and need for dialysis or hemofiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Misericordia e Dolce, Prato, Prato, Italy